CLINICAL TRIAL: NCT01594775
Title: Oxytocin, Couple Interaction and Wound Healing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KEK-ZH-NR: 2009-0063
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Oxytocin; Nasal Sprays

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- nasal spray (Active Comparator)
  Interventions: Drug: Syntocinon (Oxytocin) nasal spray
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Syntocinon (Oxytocin) nasal spray — two-times daily self-administration of nasal spray containing active substance (oxytocin) during five days after wounding.
  Arms: nasal spray
Drug: Placebo — two-times daily self-administration of nasal spray containing placebo during five days after wounding.
  Arms: Placebo

SUMMARY:
effects of intranasal oxytocin and couple interaction on wound healing.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* healthy heterosexual couples
* in a stable relationship since > 1 year

Exclusion criteria: pregnancy

* breast feeding
* heavy smoking (> 5 cigarettes/d)
* extensive skin disease
* artificial UV irradiation during < 3 months before study inclusion

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
wound size | seven days
  wound healing process within seven days after wounding

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Severin Laeuchli, MD, Principal Investigator — University Hospital Zurich, Division of Dermatology
Locations (1):
- University Hospital Zurich, Dept. of Dermatology, Zurich, Switzerland

REFERENCES:
- [Derived] Schneider E, Hernandez C, Brock R, Eckstein M, Bodenmann G, Heinrichs M, Ehlert U, Lauchli S, Ditzen B. Intranasal Oxytocin and Physical Intimacy for Dermatological Wound Healing and Neuroendocrine Stress: A Randomized Clinical Trial. JAMA Psychiatry. 2025 Nov 12:e253705. doi: 10.1001/jamapsychiatry.2025.3705. Online ahead of print. PMID 41222549
- [Derived] Aguilar-Raab C, Stoffel M, Fischer M, Eckstein M, Bodenmann G, Heinrichs M, Ehlert U, Ditzen B. Minimal couple intervention to improve psychobiological stress resilience. Br J Health Psychol. 2025 May;30(2):e12799. doi: 10.1111/bjhp.12799. PMID 40356464
- [Derived] Doerr JM, Klaus K, Troxel W, Nater UM, Bodenmann G, Heinrichs M, Ehlert U, Ditzen B. The Effect of Intranasal Oxytocin on the Association Between Couple Interaction and Sleep: A Placebo-Controlled Study. Psychosom Med. 2022 Jul-Aug 01;84(6):727-737. doi: 10.1097/PSY.0000000000001091. Epub 2022 Apr 27. PMID 35472193